CLINICAL TRIAL: NCT06880913
Title: A Phase I Dose-Escalation and Phase II Study of Nanobody-Based CD19/CD22 Tandem Dual Chimeric Antigen Receptor (CAR) T-cell Therapy in Patients With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia
Brief Title: Nanobody-Based CD19/CD22 Tandem Dual CAR-T Therapy for R/R B-ALL
Acronym: Phase I/II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Director of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHD024-001
Record Dates: First submitted 2025-03-08; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Precursor B-Cell Lymphoblastic Leukemia-Lymphoma
Keywords: R/R B-ALL
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Phase I, a traditional 3+3 dose-escalation design and determine the recommended Phase II dose; Phase II, a single-arm, open-label study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/CD22 Tandem Dual CAR-T (Experimental): Eligible patients will be treated with Nanobody-Based CD19/CD22 Tandem Dual CAR-T
  Interventions: Biological: Nanobody-Based CD19/CD22 Tandem Dual CAR-T

INTERVENTIONS:
Biological: Nanobody-Based CD19/CD22 Tandem Dual CAR-T — Phase I: Patients will receive a single infusion of autologous CD19/CD22 dual CAR-T cells at one of three dose levels (0.3 × 10⁶ cells/kg, 1.0 × 10⁶ cells/kg, or 2.0 × 10⁶ cells/kg) following fludarabine (25-30mg/m2*3d) and cyclophosphamide (250-300mg/m2*3d) (FC) lymphodepleting chemotherapy.
  Phase II: Patients will receive autologous CD19/CD22 dual CAR-T cells at the RP2D following FC lymphodepleting chemotherapy.

SUMMARY:
To evaluate the efficacy and safety of Nanobody-Based CD19/CD22 Tandem Dual Chimeric Antigen Receptor (CAR) T-cell therapy in patients with relapsed or refractory B-ALL

DETAILED DESCRIPTION:
This Phase I/II study aims to evaluate the safety, tolerability, and efficacy of Nanobody-Based CD19/CD22 Tandem Dual CAR-T-cell therapy in patients with relapsed or refractory (R/R) B-cell acute lymphoblastic leukemia (B-ALL), particularly those who have failed or relapsed after CD19- or CD22-targeted CAR-T or antibody-based immunotherapy.

In the Phase I portion of the study, a 3+3 dose-escalation design will be employed to evaluate safety and determine the optimal dose of Nanobody-Based CD5 CAR-T cells. Three dose levels will be tested: 0.3 × 10⁶ cells/kg, 1.0 × 10⁶ cells/kg, and 2.0 × 10⁶ cells/kg. The recommended Phase II dose (RP2D) will be established based on safety data, dose-limiting toxicities (DLTs), and preliminary efficacy outcomes.

The Phase II portion will then focus on evaluating the efficacy of Nanobody-Based CD19/CD22 Tandem Dual CAR-T therapy at the RP2D, with key endpoints including overall response rate (ORR), duration of response (DOR), disease-free survival (DFS), and overall survival (OS). Safety assessments, including cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS), will also be conducted throughout the study.

This study seeks to address the unmet clinical need for effective treatment options in patients with R/R B-ALL, particularly those who have exhausted prior CD19- or CD22-directed therapies.

ELIGIBILITY:
Inclusion Criteria:

The subject or their legally authorized representative (guardian) understands the study and voluntarily signs the informed consent form (ICF).

Male or female, aged 3 to 65 years at the time of signing the ICF (inclusive of the cutoff values).

Expected survival of at least 12 weeks. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at the time of signing the ICF.

At the time of signing the ICF, the patient must be diagnosed with R/R B-ALL and meet the following criteria:

1. Bone marrow morphological examination at screening shows >5% blasts in the bone marrow, and/or cerebrospinal fluid (CSF) analysis detects leukemic cells, and/or the presence of measurable extramedullary lesions, defined as:

   Any lymph node or mass with an axial diameter >1.5 cm Any extranodal lesion with an axial diameter >1.0 cm
2. Flow cytometry confirms CD19 or CD22 positivity in tumor cells from bone marrow, peripheral blood, or cerebrospinal fluid, or pathology confirms CD19 or CD22 positivity in lymph nodes/masses or extranodal lesions.

Adequate organ function, meeting the following laboratory criteria:

1. Liver function:

   Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5× upper limit of normal (ULN) Total bilirubin ≤2× ULN
2. Renal function:

Adults: Serum creatinine clearance ≥60 mL/min (using the Cockcroft-Gault formula) or creatinine ≤1.5× ULN

Children: Serum creatinine levels must not exceed the following values:

10-13 years: ≤1.2 mg/dL Males 13-16 years: ≤1.5 mg/dL Females ≥13 years: ≤1.4 mg/dL Males ≥16 years: ≤1.7 mg/dL Blood oxygen saturation (SpO₂) >92% on room air. Fertile male and female subjects of reproductive potential must agree to use effective contraception from the time of informed consent until 2 years after administration of the study drug.

Women of childbearing potential (WOCBP) include premenopausal women and those within 2 years post-menopause.

A negative blood pregnancy test is required for all female participants of childbearing potential at screening.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. History of central nervous system (CNS) diseases, including but not limited to:

   * Epilepsy
   * Paralysis
   * Aphasia
   * Stroke
   * Severe brain injury
   * Dementia
   * Parkinson's disease
   * Neuropathy
2. History of autoimmune diseases requiring systemic immunosuppressive therapy within 2 years prior to signing the ICF, including but not limited to:

   * Crohn's disease
   * Rheumatoid arthritis
   * Systemic lupus erythematosus (SLE)
   * Systemic sclerosis
   * Inflammatory bowel disease (IBD)
   * Vasculitis
   * Psoriasis
3. Presence of any uncontrolled active infection at the time of signing the ICF or within 4 weeks prior to apheresis that requires antibiotic, antiviral, or antifungal treatment.
4. Positive virological or infectious disease markers, including:

   * Hepatitis B virus (HBV): Subjects with positive HBsAg or HBcAb-positive at screening must have undetectable HBV DNA in peripheral blood to be eligible; otherwise, they should be excluded.
   * Hepatitis C virus (HCV): Subjects with positive HCV antibodies and detectable HCV RNA should be excluded.
   * Human immunodeficiency virus (HIV) antibody-positive subjects should be excluded.
   * Cytomegalovirus (CMV) DNA test-positive subjects should be excluded.
   * Epstein-Barr virus (EBV) DNA test-positive subjects should be excluded.
   * Positive serological or non-specific antibodies for Treponema pallidum (syphilis).
5. Clinically significant cardiovascular diseases, including any of the following:

   1. QTc interval ≥480 ms (Fridericia correction formula)
   2. New York Heart Association (NYHA) Class II or higher heart failure
   3. Unstable angina or acute myocardial infarction within 6 months prior to signing the ICF
   4. Left ventricular ejection fraction (LVEF) <50%
   5. Poorly controlled hypertension (as determined by the investigator)
   6. Clinically significant arrhythmias or those requiring antiarrhythmic treatment, including:

      * Persistent ventricular tachycardia
      * Ventricular fibrillation
      * Torsades de pointes
      * Complete left bundle branch block
6. History of severe hypersensitivity or allergy to any components of the study drug.
7. Receipt of any investigational drug therapy or other systemic antitumor therapy within 4 weeks before apheresis (or 5 half-lives of the drug, whichever is longer, as determined by the investigator).
8. Receipt of extensive radiotherapy within 4 weeks prior to signing the ICF, except for palliative radiotherapy for non-target lesions within 2 weeks before signing the ICF or as expected during the study.
9. Unresolved toxicity from prior antitumor therapy that has not returned to Grade 1 or baseline levels at the time of signing the ICF, except for hair loss and pigmentation (per NCI-CTCAE v5.0).
10. Requirement for systemic corticosteroids or other immunosuppressive therapy (≥10 mg/day prednisone or equivalent) within 3 days prior to apheresis or during the study period, except for:

    1. Intranasal, inhaled, or topical steroids, or localized steroid injections (e.g., intra-articular injections)
    2. Systemic corticosteroids ≤10 mg/day prednisone (or equivalent physiological dose)
    3. Steroids as prophylaxis for allergic reactions (e.g., pre-medication before contrast-enhanced CT)
    4. Steroids used for symptomatic treatment of transfusion-related reactions
11. Major surgery within 4 weeks prior to signing the ICF (excluding routine biopsy procedures) or planned major surgery during the study period.
12. History of active tuberculosis infection within 1 year prior to signing the ICF, except for subjects with a history of tuberculosis more than 1 year ago, provided that the investigator determines there is no evidence of active tuberculosis.
13. History of other primary malignancies within 5 years prior to signing the ICF, except for:

    1. Adequately treated carcinoma in situ of the cervix
    2. Localized basal cell carcinoma or squamous cell carcinoma of the skin
14. Receipt of live-attenuated or inactivated vaccines within 4 weeks before signing the ICF or planned vaccination during the screening period.
15. Any other condition or complication that, in the investigator's judgment, may affect adherence to the study protocol or make the subject unsuitable for participation.
16. Pregnancy or lactation.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Day28 after CAR-T cell infusion
  CRS and ICANS will be assessed per ASTCT (2019), while other AEs follow CTCAE v5.0. DLTs are CAR-T-related AEs (possibly, likely, or definitely related) that occur within 28 days post-infusion and meet the following criteria:
  Grade 4+ CRS, or Grade 3 CRS unresolved to ≤ Grade 2 within 7 days. Grade 3+ non-hematologic toxicity unresolved to ≤ Grade 2 within 7 days. Grade 4+ ICANS, or Grade 3 ICANS unresolved to ≤ Grade 2 within 3 days. Grade 4+ hematologic toxicity (excluding lymphopenia) lasting >28 days. Grade 3+ hypersensitivity reaction. Any unexpected toxicity requiring study discontinuation.
  Exemptions:
  Rapid hypersensitivity resolving to ≤ Grade 2 in 2 hours. Reversible Grade 3 AEs lasting ≤7 days. Transient CRS-related organ dysfunction, resolving in ≤7 days per SRC. All DLTs are reviewed by the Safety Review Committee.
Overall Response Rate (ORR) | Within 3 months after CAR-T cell infusion
  Time Frame: Within 3 months after CAR-T cell infusion Definition: ORR is defined as the proportion of patients achieving complete remission (CR), complete remission with incomplete hematologic recovery (CRi), or morphologic leukemia-free state (MLFS), as per European LeukemiaNet (ELN) 2022 criteria.
  Response Criteria (ELN 2022):
  Complete Remission (CR):
  <5% bone marrow blasts Absolute neutrophil count (ANC) ≥1.0 × 10⁹/L Platelet count ≥100 × 10⁹/L No evidence of extramedullary disease Full hematologic recovery
  Complete Remission with Incomplete Hematologic Recovery (CRi):
  <5% bone marrow blasts ANC <1.0 × 10⁹/L and/or platelet count <100 × 10⁹/L No evidence of extramedullary disease
  Morphologic Leukemia-Free State (MLFS):
  <5% bone marrow blasts No hematologic recovery required (ANC and platelet counts may remain low) No extramedullary leukemia

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | 2-year
  DFS is defined as the duration from the first confirmed complete remission (CR), complete remission with incomplete hematologic recovery (CRi), or morphologic leukemia-free state (MLFS) to the occurrence of:
  Bone marrow relapse - defined as the recurrence of ≥5% blasts in the bone marrow.
  Extramedullary relapse - defined as the recurrence of leukemia outside the bone marrow, such as in the central nervous system (CNS), lymph nodes, liver, spleen, or other organs.
  Death from any cause, whichever occurs first.
Overall Survival (OS) | 2-year
  Overall Survival (OS) is defined as the duration from the first CAR-T cell infusion to the date of death from any cause. Patients who are still alive at the time of analysis will be censored at their last known follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-jun Huang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Deparment of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided